CLINICAL TRIAL: NCT06048796
Title: Early Cessation of Sedation and TTM in Patients With a Favourable EEG After Cardiac Arrest: a Feasibility and Safety Study
Brief Title: Early Cessation of Sedation and TTM in Patients With a Favourable EEG After Cardiac Arrest
Acronym: SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: Rijnstate Hospital (Other); University of Twente (Other)
Responsible Party: Principal Investigator, Marleen Tjepkema-Cloostermans, Technical Physician Specialist, Medisch Spectrum Twente
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SELECT; NL84714.100.23 (Registry Identifier: ToetsingOnline)
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hypoxia-Ischemia, Brain; Heart Arrest
Keywords: EEG; targeted temperature management (TTM)
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Heart Arrest

STUDY DESIGN:
Intervention Model Description: A cluster randomized crossover design with two treatment arms (early cessation from sedation and TTM vs standard care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cessation of sedation and TTM (Experimental): Early cessation of sedation and targeted temperature management (TTM), with subsequent weaning from mechanical ventilation if appropriate (intervention group).
  Interventions: Other: Early cessation of sedation and TTM
- Standard Care (No Intervention): Standard care, including sedation and targeted temperature management (TTM) for at least 24-48 hours (control group).

INTERVENTIONS:
Other: Early cessation of sedation and TTM — Early cessation of sedation and TTM, with subsequent weaning from mechanical ventilation if appropriate
  Arms: Early cessation of sedation and TTM

SUMMARY:
The objective of this study is to estimate the feasibility and safety of early weaning from ICU treatment in patients after cardiac arrest and an early (< 12 h) favourable EEG pattern (indicating no or mild postanoxic encephalopathy).

DETAILED DESCRIPTION:
Comatose patients after cardiac arrest are treated on intensive care units with sedative medication, targeted temperature management (TTM), mechanical ventilation, and hemodynamic support. Despite substantial variation in the severity of the encephalopathy and even lack of unequivocal evidence of efficacy of sedation and TTM, all patients receive standard treatment. The severity of the postanoxic encephalopathy can reliably be assessed with the electroencephalogram (EEG). A continuous EEG pattern within the first 12 hours after cardiac arrest ("favorable EEG") is strongly associated with a good neurological outcome and reflects a very mild or transient encephalopathy. The investigators hypothesize that this subgroup of patients, with a favorable EEG will not benefit from prolonged sedation and TTM.

The objective of this study is to estimate the feasibility and safety of early weaning from ICU treatment in patients after cardiac arrest and an early (< 12 h) favourable EEG pattern. The study design is a cluster randomized crossover design with two treatment arms. The intervention contrast will be early cessation of sedation and TTM, with subsequent weaning from mechanical ventilation if appropriate (intervention group) vs. standard care, including sedation and TTM for at least 24-48 hours (control group). The investigators will include forty adult patients admitted to the ICU with postanoxic encephalopathy after cardiac arrest and an early (<12 hours) favorable EEG pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patients after cardiac arrest admitted to the ICU for treatment with sedation, TTM and mechanical ventilation.
* Age 18 years or older.
* Continuous EEG measurement started within 12 hours after cardiac arrest.
* Favourable EEG pattern within 12 hours after arrest, defined as a continuous background pattern (NVN, 2019; Ruijter et al., 2019).
* Possibility to stop sedative treatment within three hours after identification of a favourable EEG pattern.
* Written informed consent (deferred).

Exclusion Criteria:

* A known history of another medical condition with limited life expectancy (<6 months).
* Any progressive brain illness, such as a brain tumour or neurodegenerative disease.
* Pre-admission Glasgow Outcome Scale Extended score of 4 or lower.
* Reason other than neurological condition to continue sedation and/or ventilation.
* Follow-up impossible due to logistic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time in hours | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).

SECONDARY OUTCOMES:
Length of ICU stay | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).
Total sedation time | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).
Need for re-intubation | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).
Need for restarting sedation | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).
Number of serious adverse events (SAEs) | at 3 and 6 months
Mortality | at 30 days, 3 months and 6 months
Complications during intensive care admission | During the complete ICU admission (from admission to the ICU until discharge from the ICU, up to 30 days).
  Number of pneumonia, sepsis (according to sepsis 3 criteria), bleeding (any cause), cardiac arrhythmia (any associated with hemodynamic compromise), new cardiac arrest and thrombopenia
Neurological outcome measured at the Extended Glasgow Outcome Scale (GOSE) | at 3 and 6 months
  The CPC ranges from 1 to 8, with higher scores meaning better neurological outcome.
Neurological outcome measured at the Cerebral Performance Category (CPC) | at 3 and 6 months
  The CPC ranges from 1 to 5, with higher scores meaning worse neurological outcome.
Cognitive functioning | at 3 and 6 months
  Montreal Cognitive Assessment (MOCA) score via videoconference. The MOCA ranges from 0 to 30, with higher scores meaning better cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate hospital, Arnhem, Gelderland
  - Medisch Spectrum Twente, Enschede, Overijssel

IPD SHARING:
Plan to Share IPD: No